CLINICAL TRIAL: NCT06932419
Title: Ozone Reaction Products and Their Acute Effects on Skin Health: a Randomized Controlled Study
Brief Title: Ozone Reaction Products and Skin Health
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haidong Kan, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: FDUEH-10
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Skin Health
Keywords: Ozone reaction products; Skin health

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exposure group (Experimental): The forearm assigned to this group will be exposed to 200 ppb ozone for 2 hours.
  Interventions: Other: Ozone exposure
- Control group (Sham Comparator): The forearm assigned to this group will be exposed to clean air for 2 hours.
  Interventions: Other: Clean air exposure

INTERVENTIONS:
Other: Ozone exposure — Participants' forearms were exposed to 200 ppb ozone for 2 h at a temperature and relative humidity of 27±2°C and 45%±5%, respectively.
  Arms: Exposure group
Other: Clean air exposure — Participants' forearms were exposed to clean air for 2 h at a temperature and relative humidity of 27±2°C and 45%±5%, respectively.
  Arms: Control group

SUMMARY:
This is a randomized controlled human exposure study. Investigators aim to investigate the products of ozone-sebum reactions and their acute effects on skin health of healthy young adults.

DETAILED DESCRIPTION:
The investigators will conduct a randomized, controlled human exposure study involving 40 healthy young adults in Shanghai, China. Each participant will have both forearms simultaneously exposed-one in a clean air chamber and the other in an ozone chamber-for 2 hours. The ozone concentration at the ozone chamber inlet will be maintained at 200 ppb. The temperature and relative humidity in both chambers will be maintained at 27±2℃ and 45%±5%, respectively. Health examinations will be conducted at three time points: immediately before exposure, immediately after exposure, and 24 hours after exposure. These examinations will include skin measurements and sampling.

ELIGIBILITY:
Inclusion Criteria:

* Living in Shanghai during the study period;
* Having healthy skin conditions on both forearms.

Exclusion Criteria:

* Subjects with a history of smoking and alcohol abuse;
* Subjects with a regular use of medication and dietary supplements within 2 months prior to enrollment;
* Subjects with severe skin diseases, such as atopic dermatitis, eczema, or severe acne;
* Subjects with allergic diseases, such as allergic rhinitis, allergic asthma, or atopy, or history of allergic reactions within 2 months prior to enrollment;
* Subjects with cardiovascular diseases, such as congenital heart disease, pulmonary heart disease, or hypertension;
* Subjects with respiratory diseases, such as asthma, acute or chronic bronchitis, or pneumonia;
* Subjects with chronic diseases, such as diabetes, chronic hepatitis, or kidney disease;
* Subjects with cutaneous abnormalities on forearm, such as severe pigmentation, multiple nevus, or tattooing;
* Subjects who underwent cosmetic intervention on forearms within 2 months prior to enrollment, such as whitening treatments, UV exposure therapies, depigmentation procedures, or tanning;
* Females in pregnancy or lactation status.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Changes in chemical exposome level on the forearm skin | Immediately before exposure and immediately after exposure.
  Changes in the amount and level of chemical contaminants between ozone and clean air exposures, which will be detected using non-targeted or targeted methods.

SECONDARY OUTCOMES:
Changes in skin hydration | Immediately before exposure, immediately after exposure, and 24 hours after exposure.
  Changes in the amount of skin hydration, which will be measured by a hydration meter.
Changes in TEWL | Immediately before exposure, immediately after exposure, and 24 hours after exposure.
  Changes in transepidermal water loss on the forearm, which will be measured by an evaporimeter.
Changes in pH | Immediately before exposure, immediately after exposure, and 24 hours after exposure.
  Changes in the pH level of skin, which will be measured by a PH meter.

OTHER OUTCOMES:
Differences in skin microbiome | Immediately after exposure.
  Differences in skin microbiome between ozone exposure and clean air exposure, which will be measured using sterile swab samples.
Changes in TNF-α | Immediately before exposure and immediately after exposure.
  Changes in the level of tumour necrosis factor-α on the forearms, which will be measured using D-squame tape samples.
Changes in IL-1α | Immediately before exposure and immediately after exposure.
  Changes in the level of interleukin-1α on the forearms, which will be measured using D-squame tape samples.
Changes in pyrrolidone carboxylic acid | Immediately before exposure, and immediately after exposure.
  Changes in the amount of pyrrolidone carboxylic acid on the forearms, which will be measured using D-squame tape samples.
Changes in total protein levels of stratum corneum | Immediately before exposure, and immediately after exposure.
  Changes in the amount of total protein on forearms stratum corneum, which will be detected using D-squame tapes.
Changes in carbonyl protein | Immediately before exposure, and immediately after exposure.
  Changes in the amount of carbonyl protein on the forearms, which will be measured using D-squame tape samples.
Changes in total antioxidant capacity | Immediately before exposure, and immediately after exposure.
  Changes in the amount of total antioxidant capacity on the forearms, which will be measured using D-squame tape samples.
Changes in GSH | Immediately before exposure, and immediately after exposure.
  Changes in the level of glutathione on the forearms, which will be measured using D-squame tape samples.

CONTACTS AND LOCATIONS:
Overall Officials: Yue Niu, PhD, Study Director — Department of Environmental Health, School of Public Health, Fudan University
Locations (1):
- Department of Environmental Health, School of Public Health, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No